CLINICAL TRIAL: NCT03943758
Title: Effect of a Prepackaged Low-residue Diet on Bowel Preparation for Colonoscopy
Brief Title: a Low-residue Diet for Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Jinan Military General Hospital (Other); Wuhan TongJi Hospital (Other); Zhejiang University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Low-residue
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Colon Polyp; Colorectal Adenoma
Keywords: Bowel preparation; Polyp; adenoma
MeSH Terms: conditions — Colonic Polyps; Polyps; Adenoma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prepackaged Low-residue diet group (Experimental): The prepackaged Low-residue diet (Maifu Nutrition Technology Co. Ltd, Beijing, China). One package of the prepackaged Low-residue diet contained quantity of heat amounts to 268 kilocalories with 12.0 g of protein, 9.6 g of lipid, and 34.1 g of carbohydrate.
  Interventions: Dietary Supplement: Prepackaged Low-residue diet
- self-prepared Low-residue group (Active Comparator): Subjects in the self-prepared Low-residue diet group were instructed to follow and prepare an Low-residue diet in the day prior to colonoscopy
  Interventions: Dietary Supplement: Self-prepared Low-residue diet

INTERVENTIONS:
Dietary Supplement: Prepackaged Low-residue diet — Subjects in the prepackaged Low-residue diet group were given 6 packs (60g/pack) pre-packaged formula LRD and asked to use the formula according to individual needs prior to colonoscopy.
  Arms: prepackaged Low-residue diet group
Dietary Supplement: Self-prepared Low-residue diet — Subjects in the self-prepared Low-residue diet group were instructed to follow and prepare an Low-residue diet in the day prior to colonoscopy.
  Arms: self-prepared Low-residue group

SUMMARY:
Previous researches demonstrated that a prepackaged low-residue diet (LRD) could achieve better bowel preparation quality compared with a self-prepared LRD. However, up to now, there has been no widely acceptable standard of LRD for bowel preparation. Moreover, these prepackaged LRD adopted in previous studies mainly consisted of traditional foods without further processing. Recently, a prepackaged LRD for Special Medical Purpose was specifically designed for bowel preparation. This trail was to compare the impact of the prepackaged LRD on bowel preparation for colonoscopy with self-prepared LRD by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is between 18-65.
* Patients who have indications for screening, surveillance and diagnostic colonoscopy.
* Patients who have signed inform consent form

Exclusion Criteria:

* subjects who had known or suspected heart failure, stroke or renal failure;
* subjects who had a history of colon surgery or inflammatory bowel disease;
* subjects who Patients with had digestion or absorption dysfunction or any dietary restriction due to various reasons;
* subjects who had a history of hypersensitivity to any ingredients of laxatives or soy products;
* subjects who had high risk factors for bowel preparation such as chronic constipation, Body Mass Index (BMI) greater than 30 or BMI less than 18 Kg/m2, diabetes, spinal cord injury, or use of medications affecting bowel motility within a week;
* subjects who had participated in another interventional clinical trial in the previous 60 days;
* pregnant or lactating women and those planning to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation rate | 30 mins
  Boston Bowel Preparation Scale (BBPS) was adopted to evaluate the quality of bowel preparation. Each section of the colon (i.e. the right, the transverse, and the rectosigmoid colon) was rated (0, very poor; 1, poor; 2, good; and 3, very good). Adequate bowel of bowel preparation was defined as a total score ≥ 6 and all colon segments BBPS ≥ 2. Inadequate bowel preparation was defined as any colon segment BBPS ≤ 1.
BBPS scores of the entire colon | 30 mins
  The sum of the scores of three bowel segment.

SECONDARY OUTCOMES:
adenoma detection rate (ADR) | 30 mins
  adenoma detection rate is the number of patients with at least one adenoma, divided by the total number of patients.
preparation completion rate | 1 day
  preparation completion rate is the number of patients ingest more than 80% laxative, divided by the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan P, Gu L, Zhao S, Wang S, Ma J, Fu H, Chen Y, He S, Tian Z, Xu L, Feng Z, Li Y, Yang Z, Yang L, Wang W, Hou Q, Liu T, Li C, Tian D, Wang X, Gao Y, Shi H, Bai Y, Li Z. Prepackaged formula low-residue diet vs. self-prepared low-residue diet before colonoscopy: A multicenter randomized controlled trial. Front Med (Lausanne). 2023 Mar 24;10:1029493. doi: 10.3389/fmed.2023.1029493. eCollection 2023. PMID 37035340